CLINICAL TRIAL: NCT01077167
Title: An Open Label, Multiple Dose Study to Investigate the Pharmacokinetics of Omecamtiv Mecarbil Administered Orally to Patients With Stable Heart Failure
Brief Title: Pharmacokinetic Study of Omecamtiv Mecarbil in Heart Failure Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Study cancelled due to sponsor's decision to redesign the study
Sponsor: Cytokinetics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 20090618
Record Dates: First submitted 2010-02-25; First posted 2010-02-26 (Estimated); Last update posted 2021-07-30 (Actual); Status verified 2021-07

CONDITIONS: Heart Failure
Keywords: Omecamtiv mecarbil; pharmacokinetics
MeSH Terms: conditions — Heart Failure | interventions — omecamtiv mecarbil

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Omecamtiv mecarbil

INTERVENTIONS:
Drug: Omecamtiv mecarbil — Oral dosing twice each day or three times each day, depending on the cohort assignment, of Omecamtiv mecarbil for 8 days. Omecamtiv mecarbil comes in 2 formulations: modified release and immediate release, and the formulation given will depend on the cohort assignment.
  Other Names: AMG 423

SUMMARY:
The purpose of this trial is to obtain a pharmacokinetic profile (i.e. amount of drug in the blood over time) of Omecamtiv mecarbil in patients with stable heart failure.

DETAILED DESCRIPTION:
This study was conducted by Amgen as the IND holder, with Cytokinetics as a collaborator. Due to the termination of the collaboration agreement between Amgen and Cytokinetics in May 2021 and subsequent transfer of the omecamtiv mecarbil IND from Amgen to Cytokinetics, Cytokinetics is now listed as the sponsor.

ELIGIBILITY:
Inclusion Criteria:

* The patient has signed an Informed Consent Form/Patient Information Sheet for this study approved by the governing Institutional Review Board (IRB) or Independent Ethics Committee (IEC)
* ≥18 years old at the time of consent
* Heart failure (HF) for ≥ 3 months and New York Heart Association class II or III at enrollment
* Left ventricular ejection fraction < / = 35% by most recent echocardiogram within 3 months of enrollment. For patients with cardiac resynchronization therapy (CRT), left ventricular ejection fraction (LVEF) assessment for eligibility must be performed at least 3 months after device implantation
* Treated for HF with optimal, stable pharmacological therapy. In general, optimal treatment will include a beta-blocker and an Angiotensin Converting Enzyme (ACE) inhibitor and/or an Angiotensin Receptor Blocker (ARB) at doses shown to be efficacious in Heart Failure (HF) trials, unless not tolerated. Stable medical therapy is defined as having no new HF drug class introduced 4 weeks prior to enrollment, although doses of all drugs may be adjusted throughout the trial
* Considered to be an appropriate candidate for study enrollment as determined by the patient's clinical laboratory findings, vital signs and electrocardiograms (ECGs) within normal range, or if outside of the normal range not deemed clinically significant in the opinion of the Investigator
* For female patients only: The patient is post-menopausal (≥ 1 year) or sterilized, or if she is of childbearing potential, she is not breastfeeding, her pregnancy test is negative, she has no intention to become pregnant during the course of the study and within 1 week following the last dose of omecamtiv mecarbil, and she is using highly effective methods of birth control. Postmenopausal female is defined as 12 continuous months of spontaneous amenorrhea confirmed by a serum follicle-stimulating hormone (FSH) result > 40mIU/mL, or at least 6 weeks postsurgical bilateral oophorectomy (with or without hysterectomy) as documented in medical history (verified with an operative note, if available)
* For male patients only: Male patients agree for the duration of the study and 11 weeks after the last dose of omecamtiv mecarbil to use a condom during sexual intercourse with female partners who are of reproductive potential and to have female partners use an additional effective means of contraception (eg, diaphragm plus spermicide, or oral contraceptives) or the male subject must agree to abstain from sexual intercourse for the duration of the study and 11 weeks after the last dose of omecamtiv mecarbil.

Exclusion Criteria:

* HF hospitalization, acute coronary syndrome, myocardial infarction, percutaneous intervention coronary revascularization, transient ischemic attack or stroke, cardiac arrhythmia within 6 weeks prior to enrollment , or major surgery including thoracic or cardiac within 8 weeks prior to enrollment
* Symptoms of angina at rest or with minimal activity (Canadian Cardiovascular Society class III and IV)
* Severe aortic or mitral stenosis or clinically significant valvular heart disease that might lead to surgical correction within 12 months of enrollment
* Hypertrophic obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, or clinically significant congenital heart disease
* Refractory, end-stage, heart failure defined as subjects who are appropriate candidates in the opinion of the investigator for ventricular assist devices, continuous inotropic therapy, or hospice care
* CRT implantation within 3 months or implantable cardioverter defibrillator (ICD) within 4 weeks prior to enrollment
* Likely to receive cardiac transplant within 6 months after enrollment
* Recipient of any major organ transplant (eg, lung, liver, heart, bone marrow, renal)
* Known to be hepatitis B surface antigen, hepatitis C virus, or human immunodeficiency virus (HIV) positive, or a known diagnosis of acquired immunodeficiency syndrome
* Recent (within 3 months) history of alcohol or illicit drug abuse
* Concomitant non-cardiovascular disease that is expected to reduce life expectancy to less than 1 year
* Routinely scheduled outpatient intravenous (IV) infusions for HF (eg, inotropes, vasodilators [eg, nesiritide], diuretics) or routinely scheduled ultrafiltration
* Subjects on digoxin therapy with a steady state plasma level (approximately 6 hours post-dose) that exceeds 1.0 ng/mL at screening
* Chronic antiarrhythmic therapy, with the exception of amiodarone
* Currently taking, or has taken within 14 days prior to enrollment, a potent Cytochrome P450 3A4 (CYP3A4) inhibitor
* Currently taking, or has taken within 28 days prior to enrollment, a potent CYP3A4 inducer
* Prior treatment with omecamtiv mecarbil
* Currently enrolled in, or at least 60 days or 5 half-lives, whichever is greater, since ending participation in other investigational device or drug trial(s) or receiving other investigational agent
* Systolic blood pressure > 150 mm Hg or < 80 mm Hg, or diastolic blood pressure > 95 mm Hg, assessed on two separate occasions prior to enrollment
* Supine heart rate ≥ 100 beats per minute after 5 minutes of rest or an untreated symptomatic bradyarrhythmia within 1 month prior to enrollment
* Troponin I at screening > upper limit of normal (ULN)
* Total bilirubin ≥ 1.5 times ULN, or an Alanine transaminase (ALT) or Aspartate transaminase (AST) ≥ 3 times ULN
* Estimated glomerular filtration rate (GFR) ≤ 30 ml/min/1.73 m2 calculated by the Modification of Diet in Renal Disease (MDRD) equation
* In the opinion of the Investigator, a condition that compromises the ability of the subject to give written informed consent or to comply with study procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-07; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetic profile of oral formulations of Omecamtiv mecarbil following the morning dose on Days 7 and 8 | Following 8 Days of dosing

SECONDARY OUTCOMES:
Safety and tolerability of oral formulations of Omecamtiv mecarbil at steady state | 14 Days

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com